CLINICAL TRIAL: NCT06278441
Title: Assistant Prof. Bayburt University Faculty of Health Science Department of Nursing/Pediatric Nursing
Brief Title: The Effect of White Noise and Kangaroo Care Practices on Stress Parameters in Newborns With Heel Lancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Zila Özlem KIRBAŞ, Assistant Prof., Bayburt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Zila Özlem KIRBAŞ
Record Dates: First submitted 2024-02-12; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Healthy Newborns

STUDY DESIGN:
Intervention Model Description: This study is parallel-group, randomized controlled.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding could not be done for the participants, and the two researchers who collected the data, but the statistician and two other researchers who analyzed the results were unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White noise group (Experimental): After the newborns in the WNG group were taken to the blood collection department, white noise (55 dB) was played through a speaker standing 1 meter away from the newborn. The sound level was adjusted to 55 dB with a decibel meter. A heel lancing was performed after the newborn started listening to white noise and calmed down.
  Interventions: Other: Kangaroo care and White noise
- Kangaroo care group (Experimental): Kangaroo care was started 15 minutes before heel lancing for newborns included in KCG, and heel lancing was performed.
  Interventions: Other: Kangaroo care and White noise
- Control group (No Intervention): Control group newborns underwent routine heel lancing, and no intervention was performed.

INTERVENTIONS:
Other: Kangaroo care and White noise — CG newborns underwent routine heel lancing, and no intervention was performed.
  Arms: Kangaroo care group; White noise group

SUMMARY:
Aim: It is an examination of the effects of white noise and kangaroo care on some physiological parameters (pulse, saturation, crying duration) and stress markers (cortisol and glucose-regulated protein 78 (GRP78)) in heel lancing in newborns.

Methods: In this parallel-group, randomized controlled study, healthy newborns with a gestational age of ≥37 weeks, birth weight of >2500 g, and an Apgar score of ≥8 at the 1st minute and 5th minute were included. White noise and kangaroo care were applied to newborns in the intervention groups for heel lancing.

Results: Ninety newborns were randomized into three groups (30 in each group). A statistically significant difference was determined between the median values of total crying time according to groups (p<0.001). A statistically significant difference was determined between the median values of pulse measurements according to the interaction of group and time (p<0.001). A statistically significant difference was determined between the median values of saturation measurements according to groups (p=0.001). A statistically significant difference was determined between the mean values of cortisol and GRP78 measurements according to the group and time interaction (p<0.001).

Conclusion: It was concluded that white noise and kangaroo care help reduce newborns' stress in the case of heel lancing.

DETAILED DESCRIPTION:
This study aimed to examine the effects of white noise and kangaroo care during heel lancing in newborns on some physiological parameters (pulse, saturation, crying duration) and stress markers (cortisol and GRP78).

Study Design The study was carried out with a randomized controlled experimental design. The research was conducted in the gynecology service of a hospital between January and September 2023. In Türkiye, metabolic screenings are carried out in hospitals within the first 36-72 hours after birth, before the newborn is discharged, and in Family Health centers on the 5th day. The reason why we chose the sample group from the hospital is to both monitor physiological parameters appropriately and minimize sample loss. There are 5 neonatal nurses and 3 pediatricians working in the hospital's gynecology service. The Bayburt University Ethics Committee (2022/334) approved the study.

Participants All babies (N = 90) were randomly divided into three groups (Figure 1: Consort Flow Diagram) using a computer program (http://www.randomizer.org) and the first participants were selected and assigned by lottery method (White noise group (WNG) (1), Kangaroo care group (KCG) (2), Control group (CG) (3)). After the initial assignments were made, newborns were assigned to groups according to the numbers given by random.

Data collection tools Data; "Mother and Baby Introductory Information Form (mother's age, educational status, and several children, mode of birth and newborn's Apgar score, gestational age, gender, birth weight, and height)," "Newborn Follow-up Form (crying duration, pulse (heart rate)" and oxygen saturation before, during and after the procedure; for recording stress saliva biomarker (cortisol, GRP78) levels before and after the procedure)", "Portable Monitor," "Stopwatch (Apple Watch/JAPAN)," "Portable speaker," "Decibel" measurement device (Benetech GM1351/TURKIYE", "Orhan Osman's Colic album - Don't Let Your Baby Cry 2 (Utilizing the sounds inside the uterus in Dr. Harvey Karp's album "The Happiest Baby" and combining these sounds with his compositions, 'Colic' album)," "Salimetrics SalivaBio Infant's Swab (SIS)" (It is a material used to collect the saliva of babies and newborns under six months of age. Its features are that saliva is obtained by keeping it under the tongue and in the corners of the mouth for 60-90 seconds and placed in the storage tube.) gathered.

Procedure and interventions Before the heel lancing, the mothers of newborns who met the sampling criteria were informed about the research, their written and verbal consent was obtained, and their information was recorded on the mother and baby descriptive form before the procedure. With standardization in the procedure technique, the environmental factors to which the newborns were exposed were ensured to be the same in all groups (needle tip (21 gauge, temperature (24-25 °C), light, and noise). Half an hour before the heel lancing, the newborns were fed, and their diapers were changed. It was ensured that the newborns were not exposed to painful procedures before the procedure. Crying times were monitored with a stopwatch from the beginning of the procedure until the end of the procedure and recorded in the follow-up form. Physiological parameters (pulse, O2 saturation) were monitored with a portable monitor device before, during, and after the procedure and recorded in the follow-up form. Saliva samples were collected just before the heel lancing and 20 minutes after the procedure. Necessary white noise and kangaroo care protocols were initiated before the heel lancing. For the interventions to be performed on all groups, the procedure was applied to newborns between 7:00 and 10:00 in the morning. The same neonatal nurse performed the heel lancing in each group. The researchers conducted applications, monitoring of physiological parameters, and saliva collection. Kangaroo care was started 15 minutes before heel lancing for newborns included in KCG, and heel lancing was performed. The application was carried out according to WHO's (2003) kangaroo care guide.16 After the newborns in the WNG group were taken to the blood collection department, white noise (55 dB) was played through a speaker standing 1 meter away from the newborn. The sound level was adjusted to 55 dB with a decibel meter. A heel lancing was performed after the newborn started listening to white noise and calmed down. CG newborns underwent routine heel lancing, and no intervention was performed. Due to the nature of the intervention, blinding could not be done for the participants, and the two researchers who collected the data, but the statistician and two other researchers who analyzed the results were unaware of group allocation.

Saliva collection and measurement To collect samples, the research team held one end of the saliva swab (Salimetrics® SalivaBio Infant Swab, Carlsbad, CA) and placed the other end of the swab against the newborn's buccal mucosa or sublingually to absorb saliva. Immediately after saliva collection, the swabs were labeled in storage tubes.17 The saliva samples obtained as a result of the study were transferred to Eppendorf tubes and centrifuged at 1500 g for 15 minutes in a refrigerated centrifuge (NF 1200R, NUVE, Ankara, TURKIYE) in the laboratory and then stored at -30°C until cortisol hormone and GRP78 analyzes were performed on the saliva samples. The commercial kits used in measurements are human-specific and for cortisol level (BT LAB, Cat.No E 1 003Hu, CHINA); (SinoGeneClon, ELISA Kit Product code: SG-20252, CHINA) was used for GRP78 level measurement.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥37 weeks
* Birth weight >2500 g
* Apgar score ≥8 at the 1st minute and 5th minute
* No anatomical or physiological problems
* No congenital or acquired hearing-related disease
* Newborns were born who had no malformations
* No family members with hearing loss that started in childhood

Exclusion Criteria:

* Infants receiving sedative medications
* Any evidence of dysfunction of the hypothalamic-pituitary-adrenal axis

Ages: 32 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Ninety newborns were randomized into three groups (30 in each group). | 45-60 minutes
  A statistically significant difference was determined between the median values of total crying time according to groups (p<0.001). A statistically significant difference was determined between the median values of pulse measurements according to the interaction of group and time (p<0.001). A statistically significant difference was determined between the median values of saturation measurements according to groups (p=0.001). A statistically significant difference was determined between the mean values of cortisol and GRP78 measurements according to the group and time interaction (p<0.001).

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt University, Bayburt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirbas ZO, OdabasI Aktas E, Bayraktar B, Ozkan H. Effect of kangaroo mother care and white noise on physiological-stress parameters in heel lancing: randomized controlled study. BMC Pediatr. 2024 Sep 6;24(1):568. doi: 10.1186/s12887-024-05033-1. PMID 39243091